CLINICAL TRIAL: NCT02442713
Title: A Baseline Controlled Study With Fluvoxamine to Evaluate the Effect on Polysonogram in Depressed Patients With Insomnia
Brief Title: The Effect of Fluvoxamine on Polysonogram in Depressed Patients With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang Dong Provincial Mental Health Institute (Other)
Responsible Party: Principal Investigator, Bin Zhang, Professor, Guang Dong Provincial Mental Health Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUVD002
Record Dates: First submitted 2015-04-28; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Depression
Keywords: Polysomnograph; fluvoxamine
MeSH Terms: conditions — Depression | interventions — Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluvoxamine (Experimental): fluvoxamine: 50-300mg/day
  Interventions: Drug: fluvoxamine

INTERVENTIONS:
Drug: fluvoxamine — fluvoxamine: 50-300mg/day
  Other Names: Luvox

SUMMARY:
Major depressive disorder is associated with several sleep Polysomnograph (PSG) findings: (1) impaired sleep continuity; (2) non-REM (NREM) changes; and (3) enhanced rapid eye movement (REM) sleep. The first two patterns are common in other psychiatric disorders, while the REM pattern is very characteristic in depression, so the phase-advance theory was accepted by most of psychiatrists. Many researchers have focused on the biological rhythm to investigate the etiological and pathophysiology of depression, and they think depression can be cured if its sleep abnormality is ameliorated.

It is well known that most of antidepressants treat depression through 5-hydroxytryptamine (5-HT) neurons. 5-HT also affects the regulation of the sleep-wake cycle and the sleep microarchitecture. Many all-night PSG studies have shown tricyclic antidepressants can ameliorate the sleep architecture abnormality in depression by producing rapid suppression of REM sleep.

Compared to TCAs, SSRIs are generally less sedating because of its high selectivity for serotonin receptors. On the other hand, it is known that, although all of SSRIs mainly increase the extracellular serotonin level by inhibiting serotonin transport in the presynaptic neuron, each SSRI has its unique pharmacological characteristics. For example, it was reported by accumulating researches that the serum melatonin level increased markedly after ingestion of fluvoxamine. The mechanism behind this effect is unknown, but one possibility is increased melatonin synthesis, caused by effects on serotonin, which is a melatonin precursor. Another possibility is that fluvoxamine inhibits the metabolism of melatonin in the liver.

Thus, the property of fluvoxamine to increase serum melatonin level, or even recover the circadian rhythm of melatonin in depressed patients, might improve the clinical outcome by improving the sleep quality and quantity. By now, the changes of sleep architecture in fluvoxamine treatment were assessed by only three clinical trials, and their results were contradictive. This discrepancy might be due to the small sample size and different study design, such as clinical trial duration. Moreover, two of three researches applied home-based PSG assessment, which might have distorted the results of sleep architecture to some extent. Thus, the effects of fluvoxamine on sleep architecture need to be clarified by more clinical trials with standard PSG assessment.

DETAILED DESCRIPTION:
This study is aimed to evaluate the effect of fluvoxamine on polysomnographic (PSG) variables and clinical improvement in the treatment of depressive patients with insomnia.

This is an 8-week open-label study. All patients are required to meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) [48 criteria for MDD, single or recurrent type, with moderate-to-high level of illness severity, as evidenced by a 17-item Hamilton Rating Scale for Depression (HRSD) score >17 [49, 50]. Furthermore, these depressed patients should be suffering insomnia, which was determined by the total score of sleep disturbance factor in HRSD >3 (items 4, 5, and 6; score range, 0-6).

Before any procedure of the study, the patient would be explained in detail about the potential risk and benefit in this study with a signed informed consent form (ICF). Patients can discontinue the study at any time after informed consent. Also, this study should be approved by Independent Ethics Committee (IEC) of Guang Dong Mental Health Center and compliance with the content of the declaration of Helsinki.

After 7-day wash-out period and 2 nights PSG (the first night as adaptive and the second night as baseline), 30 depressive patients were administered by fluvoxamine as 50 mg/day in the 1st day. The dosage of fluvoxamine would be titrated during the 8-week treatment, and the maximum was lower than 300 mg/day. The primary endpoints were the changes of PSG variables from baseline to the 56th Day. The secondary endpoints were the changes of subjective sleep quality and clinical performance from baseline to the 56th Day. Their sleep quality was evaluated with Epworth Sleepiness Scale (ESS) and Pittsburgh Sleep Quality Index (PSQI), and their clinical performance was evaluated with HRSD and Clinical Globe Impression (CGI).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfil all of the following criteria:

1. Male or female, ≥18 years and ≤65 years old
2. Major depressive disorder patients with insomnia (diagnosed with DSM-IV, HRSD total score >17 and total score of sleep disturbance factor in HRSD (items 4, 5, and 6; score range, 0-6)>3)
3. Patients who are able to understand and comply with the requirements of the study
4. Provision of written informed consent

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Any contraindication or caution of fluvoxamine according to Chinese label
2. Any DSM-IV Axis I disorder, except for major depressive disorder
3. Being currently treated or having been treated with fluvoxamine or other antidepressants within 4 weeks prior to entering the study
4. Participation to this study or another trial within 4 weeks prior to entering the study
5. Other sleeping disorder such as apnoea, Periodic Leg Movement in Sleep and narcolepsy
6. Pregnancy or lactation
7. Substance or alcohol dependence or any drug abuse.
8. Other conditions at Investigator's discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The change of sleep during Fluvoxamine treatment | 56 days
  by comparing the percentages of Rapid Eye Movement (REM) on the 1st, 14th, 28th and 56th day.

SECONDARY OUTCOMES:
The change of Slow Wave sleep (SWS) during Fluvoxamine treatment | 56 days
  by comparing the percentages of Slow Wave sleep (SWS) on the 1st, 14th, 28th and 56th day.
The change of sleep efficiency during Fluvoxamine treatment | 56 days
  by comparing the sleep efficiency on the 1st, 14th, 28th and 56th day.
Clinical improvement during Fluvoxamine treatment | 56 days
  by comparing scores of Hamilton Rating Scale for Depression (HRSD) on the 1st, 14th, 28th and 56th day.

CONTACTS AND LOCATIONS:
Overall Officials: 86-20-81888553 Zhang, M.D&Ph.D, Principal Investigator — Guang Dong Provincial Mental Health Institute
Locations (1):
- Guangdong Provincial Mental Health Institute, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Hao Y, Hu Y, Wang H, Paudel D, Xu Y, Zhang B. The Effect Of Fluvoxamine On Sleep Architecture Of Depressed Patients With Insomnia: An 8-Week, Open-Label, Baseline-Controlled Study. Nat Sci Sleep. 2019 Nov 4;11:291-300. doi: 10.2147/NSS.S220947. eCollection 2019. PMID 31807102